CLINICAL TRIAL: NCT01697683
Title: Probiotic Therapy for the Reversal of Bacterial Vaginosis in Pregnancy
Acronym: ProVIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0005-A
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Pregnant Women Who Test Positive for Bacterial Vaginosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic Rhamnosus Lactobacilli (Active Comparator)
  Interventions: Drug: Probiotic Lactobacilli
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic Lactobacilli — Two capsules per day containing either probiotic lactobacilli or placebo for 12 weeks
  Arms: Probiotic Rhamnosus Lactobacilli
Drug: Placebo
  Arms: Sugar pill

SUMMARY:
This study will add to the current knowledge and literature on the ability of an oral lactobacilli preparation to return the vaginal flora to a normal state in pregnant women. The results will potentially serve as the basis for a multi-centre Phase III randomized clinical trial to determine the efficacy of this treatment in preventing preterm birth.

DETAILED DESCRIPTION:
Preterm birth continues to provide the greatest challenge in perinatal health care in the developed world. It is a syndrome involving multiple causes and arises from a number of social, psychological, and biological determinants. It has been estimated that intrauterine infection accounts for at least 25-40% of spontaneous preterm births, with infection being the primary cause of extreme prematurity. Because infection-mediated preterm delivery mainly occurs in younger gestational ages (less than 28 weeks), these extremely premature babies not only have the risks associated with being born early, but are also likely to have severe morbidities associated with infection. Bacterial vaginosis (BV) is defined as a loss or significant depletion of lactobacilli coupled with an overgrowth of pathogenic bacteria and an increase in vaginal pH (>4.5). BV is common and occurs in 20% of the general female population, often without symptoms and is associated with a 40% increased risk of preterm birth. The clinical finding that lactobacilli is the dominant microbe in the vagina of women with a healthy pregnancy and full term delivery, supports the association of this species with a healthy pregnancy. BV is associated with an elevation of cervico-vaginal pro-inflammatory cytokines including IL-1β and IL-8 that are also associated with preterm labour; initiating the inflammatory cascade of events involved in labour may be the mechanism by which BV triggers preterm birth. However, not all women with BV will deliver preterm suggesting that variations in genetic susceptibility may underlie the host response to the presence of BV and the risk for preterm birth. Antibiotic therapy is the current treatment for BV, but the extent to which antibiotics can prevent preterm birth in women with BV remains somewhat uncertain, with conflicting results published in the literature. The apparent ineffective nature of antibiotic therapy, perhaps due to a lack of regrowth of lactobacilli following treatment, and the possibility that the pathogens have already induced inflammatory processes that will eventually induce preterm birth, emphasizes the need to continue to investigate the role of microbes during pregnancy. Probiotics have been suggested as an alternative to antibiotic therapy in restoring vaginal lactobacilli and reversing BV. The study seeks to determine whether Lactobacillus rhamnosus, GR-1 and Lactobacillus reuteri, RC-14 when administered to pregnant women diagnosed with bacterial vaginosis or intermediate flora will reverse the condition leading to a decrease in the inflammatory mediators involved in the cascade of infection/inflammation-mediated preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women prior to 17 weeks gestation
* singleton pregnancy
* over 18 years of age
* able to provide informed consent

Exclusion Criteria:

* multifetal pregnancies (twins, triplets, etc)
* fetal complications (congenital anomaly, chromosomal abnormality)
* maternal history of previous preterm birth or second trimester loss
* significant maternal medical or surgical complications (eg. hypertension, diabetes)
* less than 18 years of age
* unable to provide informed consent
* HIV Positive
* Immuno-compromised

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Microbial DNA profile | At 28 and at 35 weeks gestation
  A change in the Vaginal Microbial DNA profile

SECONDARY OUTCOMES:
Microbial function | At 28 and at 35 weeks gestation
  A change in microbial function as measured by RNA transcriptomics

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bocking, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada